CLINICAL TRIAL: NCT02332473
Title: A Prospective Phase 2 Clinical Trial to Assess the Efficacy and Safety of Combination of Peginterferon Alfa-2b (40kD, Y-shape) and GM-CSF in Chronic Hepatitis Patients.
Brief Title: A Prospective Study of Combination of Peginterferon Alfa-2b (40kD, Y-shape) and GM-CSF in Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1405IFN
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b; Colony-Stimulating Factors; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Ypeginterferon alfa-2b,sc. Qw. 48 weeks.
  Interventions: Drug: Ypeginterferon alfa-2b
- Arm B (Experimental): Ypeginterferon alfa-2b,sc. Qw. 48 weeks. Granulocyte-macrophage colony stimulating factor,sc.qd, the first three day of every 28 days, starting from interferon treatment week 13.
  Interventions: Drug: Ypeginterferon alfa-2b; Drug: Granulocyte-macrophage colony stimulating factor

INTERVENTIONS:
Drug: Ypeginterferon alfa-2b
  Other Names: peginterferon alfa-2b
Drug: Granulocyte-macrophage colony stimulating factor
  Other Names: GM-CSF
  Arms: Arm B

SUMMARY:
This study is a multi-center, randomized, prospective open-label study to assess the efficacy and safety of combination of peginterferon alfa-2b (40kD, Y-shape) and GM-CSF in interferon-naïve chronic hepatitis B patients with HBeAg positive. Patients were randomized to one of the 2 groups to receive different antiviral treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18yrs≤age≤65yrs.
* 17≤BMI(body mass index)≤28.
* HBsAg positive≥6 months.
* Serum HBV DNA≥20,000IU/ml, HBsAg positive and HBeAg positive at screening.
* 2ULN≤ALT≤10ULN(ULN=upper limit of normal) at screening.
* Pregnancy test must be negative for female patients of childbearing potential. All patients take effective birth control measures during treatment and 6 months after the treatment.
* Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Pregnant or lactating females
* Interferon treatment history, or using nucleos(t)ide analogues for chronic hepatitis B treatment within the previous 6 months, or any evidence of nucleosi(t)ide analogues resistance .
* Receiving strong immunomodulatory agents (e.g., steroids, thymosin) for more than two weeks 6 months prior to screening.
* Receiving hepatotoxicity agents (e.g., aczone, erythromycin, fluconazole, ketoconazole, rifampicin) for more than two weeks 6 months prior to screening.
* Co-infected with active hepatitis A, hepatitis C, hepatitis D, and/or human immunodeficiency virus (HIV).
* History or evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., autoimmune hepatitis, alcoholic liver disease, toxin exposures.
* Suffering from any other acute or chronic infectious disease.
* Mental disorder or physical disability, or family history of neurological and psychiatric disorders.
* Neutrophil count <1500 cells/mm3, or platelet count <90000 cells/mm3 at screening.
* Child-Pugh≥B, or other evidence of liver decompensation (e.g. serum albumin<35g/L , prothrombin time>3 seconds prolonged, serum bilirubin>2ULN, prothrombin activity <60%, history of liver decompensation).
* Serum creatinine level >ULN in screening period.
* Serum creatine kinase level >2ULN except for physiological factors (e.g., exercise).
* AFP>100ng/L. If 50ng/L<AFP<100ng/L at screening, retest 2 weeks later, and if AFP <50ng/L can enrolled, vs, excluded.
* Hepatocarcinoma or suffering from any other malignant tumor.
* Autoimmune disease(e.g., psoriasis, systemic lupus erythematosus).
* Moderate or severe hypertension, or mild hypertension without well controlled.
* With not well- controlled endocrine disease (e.g., thyroid dysfunction, diabetes mellitus).
* Drug abusing, or alcoholism.
* HBeAb positive or HBsAb positive at screening.
* Allergic to interferon, or GM-CSF, or any fragment of the study drug.
* Other conditions which in the opinion of the investigator precluding enrollment into the study(e.g., low compliance).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Percentage of HBeAg seroconversion at the end of treatment | week 48

SECONDARY OUTCOMES:
Percentage of HBsAg undetectable and seroconversion at the end of treatment | week 48
Percentage of HBeAg undetectable and seroconversion at week 12, 24, 36 and 48 | week 12, 24, 36 and 48
Change of HBsAg and HBeAg from baseline at week 12, 24, 36, and 48 | week 12, 24, 36, and 48
Change of HBV DNA from baseline and percentage of HBV DNA undetectable at week 12, 24, 36, and 48 | treatment week 12, 24, 36, and 48
Percentage of ALT normalization at week 24, 36 and 48 | week 24 ,36 and 48

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hosopital, Beijing, Beijing Municipality
  - Fuzhou Infectious Disease Hospital, Fuzhou, Fujian
  - Xiamen Hospital of T.C.M, Xiamen, Fujian
  - Nanfang Hospital, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Huazhong University of Science & Technology, Wuhan, Hubei
  - Xiangya Second Hospital, Central-south University, Changsha, Hunan
  - Shenyang Sixed People's Hospital, Shenyang, Liaoning
  - Ruijing Hospital, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xi’an, Shanxi
  - First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang